CLINICAL TRIAL: NCT03722940
Title: Combination of Magnesium Sulphate With Total Intravenous Anesthesia Optimized Surgical Field in Pediatric Cochlear Implant Surgery
Brief Title: Role of Magnesium in Pediatric Cochlear Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wahba bakhet (Other)
Collaborators: Bahteem Specialized Hospital (Other)
Responsible Party: Sponsor-Investigator, Wahba bakhet, Lectrure of anesthesia, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Bahtem WBAKHET
Record Dates: First submitted 2018-10-19; First posted 2018-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulphate (Active Comparator): Group M
  Interventions: Drug: Magnesium sulphate
- Na CL 0.9% (Placebo Comparator): group C
  Interventions: Other: Na CL 0.9%

INTERVENTIONS:
Drug: Magnesium sulphate — Before induction of anesthesia; children in group M received an iv bolus dose of magnesium sulfate (Magnesium sulfate ampoule 1 gm/10 ml, Eipico, Egypt) 40 mg Kg-1 over 5 minutes followed by 15 mg Kg-1 h-1 ivi until the start of skin closure.
  Other Names: MGSO4
  Arms: Magnesium sulphate
Other: Na CL 0.9% — Before induction of anesthesia; children in group C equivalent volumes of Na Cl 0.9% over the same period instead of magnesium sulphate.
  Other Names: isotonic saline solution
  Arms: Na CL 0.9%

SUMMARY:
To determine the efficiency of addition of magnesium sulfate to total intravenous anesthesia (TIVA) in optimizing the surgical field during pediatric cochlear implant surgery. Also its effects on the intraoperative evoked stapedial reflex thresholds (ESRT) and the intraoperative anesthetic requirements were evaluated.

DETAILED DESCRIPTION:
Sixty-six ASA I and II children (1-6 years) undergoing cochlear implantation under general anesthesia were enrolled in this double blind, randomized study. Children were randomly allocated into two equal groups. Children in Group M (magnesium sulphate group) received an iv bolus dose of magnesium sulfate 40 mg Kg-1 over 5 minutes before induction of anesthesia followed by 15mg Kg-1 h-1 infusion until the start of skin closure. Children in Group C (Control group) received equivalent volumes of isotonic saline solution over the same period instead of magnesium sulphate. Haemodynamic variables, quality of surgical field, ESRT and the intraoperative anesthetic requirements were recorded

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II children

Exclusion Criteria:

* uncontrolled hypertension,
* diabetes mellitus,
* liver disease,
* kidney disease,
* heart disease,
* allergy to magnesium sulphate,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Quality of surgical field | at the end of the surgey
  using Fromme's-Boezaart scale (0 to 5). A score of ≤ 2 was considered to be optimal

SECONDARY OUTCOMES:
The operative time | Intraoperative
  Minutes
The anesthesia time. | Intraoperative
  Minutes
ESRT responses | After insertion of the electrode and after reversal of any residual muscle relaxant (TOF response > 0.9),
  the surgeon assessed ESRT response at the basal, middle, and apical areas of the electrode array by visual monitoring of the stapedius muscle using direct microscopic examination
Heart rate | baseline, after surgical incision, Hypotensive period, after LMA removal and at recovery room admission.
  beats per minute
Mean arterial blood pressure | Intraoperative
  mm Hg
Anesthetic consumption | Intraoperative
  propofol and fentanyl requirement after the bolus

IPD SHARING:
Plan to Share IPD: Undecided